CLINICAL TRIAL: NCT01212588
Title: Preliminary, Double Blind, Placebo Controlled Trial of the Effect of Glucocorticoid Receptor Antagonist Treatment on Biologic and Symptom Outcomes in Patients With Borderline Personality Disorder and Histories of Childhood Abuse
Brief Title: Preliminary Trial of the Effect of Glucocorticoid Receptor Antagonist on Borderline Personality Disorder (BPD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Alan Breier, Psychiatrist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1011002977
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Borderline Personality Disorder
Keywords: BPD; Borderline; personality disorder; mifepristone
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifepristone (Experimental): Mifepristone 600mg once daily x 7 days
  Interventions: Drug: mifepristone
- Placebo (Placebo Comparator): Matching placebo tablets one daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mifepristone — Mifepristone 600mg (3x200mg tablets) once daily for seven days
  Arms: Mifepristone
Drug: Placebo — 3 tablets once daily for seven days
  Arms: Placebo

SUMMARY:
Participants will be randomized to either Mifepristone 600mg once daily for seven days or Placebo tablet once daily for seven days. Rating scales, vital signs, cortisol levels will be collected for evaluation.

DETAILED DESCRIPTION:
Mifepristone is an antagonist of type II glucocorticoid (GR-II) receptors, which has shown safety, efficacy, and good tolerability in the treatment of psychotic major depression (PMD). Like BPD, Hypothalamic-pituitary-adrenal (HPA) axis hyper-responsiveness appears to play a role in PMD pathophysiology. Belanoff et al. (2002) hypothesized that mifepristone causes a normalizing "resetting" of HPA axis rhythm, accounting for its efficacy in PMD. Mifepristone produces a marked (2- to 3- fold) compensatory increase in central cortisol levels via its antagonism of GR-II receptors. This consequent central cortisol elevation may then be able to counteract abnormally heightened corticotrophin-releasing hormone (CRH) activity via enhanced negative feedback mechanisms.

This is a proof of principle study of mifepristone in the treatment of individuals with BPD and histories of childhood abuse, which aims to translate neurobiological research concerning HPA axis abnormalities in BPD into a novel clinical intervention for patients. This project will also explore an innovative approach to the structure of pharmacotherapy for BPD. Specifically, we will employ the circumscribed (finite) drug administration period used in prior studies of mifepristone in neuropsychiatric illness, which differs from the current clinical practice of indefinite daily usage of medications. We hypothesize that mifepristone will beneficially impact stress response neurobiology and consequently ameliorate associated BPD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age at study entry
* Female or Male
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of borderline personality disorder (confirmed by SCID II) with history of abuse prior to the age of 18.
* Able to provide informed consent
* Inpatient or outpatient
* Clinical stability as defined by:

  * Subjects must not have experienced an exacerbation of their illness within 4 weeks prior to randomization, leading to an intensification of psychiatric care in the opinion of the principal investigator. Examples of intensification of care include, but are not limited to: inpatient hospitalization, day/partial hospitalization, outpatient crisis management, or psychiatric treatment in an emergency room AND
  * Psychotropic treatment stability for at least 2 weeks prior to randomization (no change in dosing or addition of any new psychotropic medication)
* Female subjects of childbearing potential must test negative for pregnancy at screening visit and agree to use the double-barrier method, as defined by 2 physical barriers such as a condom, diaphragm, or cervical occlusive cap, coupled with an additional barrier such as spermicidal foam, gel, film, cream or suppository for the duration of the study. Subjects having undergone a hysterectomy or bilateral oophorectomy or other form of female sterilization or patients having been medically confirmed to be post-menopausal, would not require any other method of contraception.
* Minimum severity of a total score > 3 on the The Clinical Global Impression severity (CGI-S)
* Must agree not to consume tonic water and grapefruit or grapefruit product for 3 days prior to beginning medication and until the final study visit

Exclusion Criteria:

* DSM-IV TR diagnosis of (confirmed by SCID) schizophrenia or a related psychotic disorder, bipolar I disorder, or dementia
* Subjects who are considered prisoners per the Indiana University Standard Operating Procedures for Research Involving Human Subjects.
* Subjects with current acute, serious, or unstable medical conditions, including, but not limited to: inadequately controlled diabetes, asthma, Chronic obstructive pulmonary disease (COPD), severe hypertriglyceridemia, recent cerebrovascular accidents, acute systemic infection or immunologic disease, unstable cardiovascular disorders, malnutrition, renal gastroenterologic, respiratory, endocrinologic (particularly illnesses related to the HPA-axis, e.g., Cushing's Syndrome), neurologic, hematologic, or infectious diseases
* Clinically significant electrocardiogram (ECG) abnormality prior to randomization including: subjects with a corrected QT interval (Bazett's; QTcB) >470 msec prior to randomization (based on the cardiologist overread). Repeat ECGs will be conducted at the discretion of the principal investigator or medical designee
* Use of any exclusionary medications listed in the protocol Attachment 2: Concomitant Medications
* Pregnant or lactating women or women who plan to become pregnant or will be lactating within one month after cessation of study medication
* Known Intelligence quotient (IQ) <70 based on medical history
* Currently using an intrauterine device (IUD) (females only)
* History of treatment with mifepristone or any mifepristone-containing medication at any time
* Known history of (1) Hepatitis C virus antibody, (2) Hepatitis B surface antigen (HBsAg) with or without positive Hepatitis B core total antibody, or (3) HIV 1 or 2 antibodies
* Subjects with moderate to severe renal impairment as defined by creatinine clearance (CrCl) < 60 ml/min (measured by the Cockcroft-Gault equation) at screening
* Subjects with hepatic impairment as defined by liver transaminases or total bilirubin > 3 × upper limit of normal (ULN)
* Subjects considered a high risk for suicidal acts, as determined by the principal investigator.
* Subjects who have participated in a clinical trial with any pharmacological treatment intervention for which they received study-related medication in the 4 weeks prior to screening OR Subjects currently receiving treatment (within 1 dosing interval plus 4 weeks) with an investigational depot formulation of an antipsychotic medication
* Subjects who demonstrate overtly aggressive behavior or who are deemed to pose a homicidal risk in the principal investigator's opinion
* Psychosocial treatment changes 14 days prior to randomization
* History of unexplained vaginal bleeding, endometrial hyperplasia with atypia, or endometrial carcinoma

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Larue D Carter Memorial Hospital, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mifepristone | Placebo
Started | 10 | 12
Completed | 9 | 10
Not Completed | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone | Placebo | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.90 (11.75) | 33.42 (10.33) | 36.82 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Rapid Symptom Change
Description: To evaluate whether mifepristone will produce rapid symptom change after seven days of active treatment, as measured by Borderline Personality Disorder Severity Index (BPDSI) total score. The BPDSI is a semi-structured clinical interview assessing the frequency and severity of manifestations of Borderline Personality Disorder (BPD) during a circumscribed period of the previous 7 days. The BPDSI measures 9 symptoms associated with BPD on a Likert scale ranging from 0-7 (0 = never; 7 = daily). Each symptom measure produces a mean score ranging from 0-7, with a higher score indicating more prevalent symptoms. A total score is then calculated using the summed symptom mean scores, ranging from 0-63, with a higher score indicating more prevalent symptoms.
Time Frame: Baseline to 7 days of study medication
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  BPDSI Total Score after 7 days of medication | 13.5 (7.93) | 9.45 (4.24)
  BPDSI Total Score at Baseline | 17.99 (6.65) | 13.66 (7.72)

2. Primary Outcome: Durable Symptom Change
Description: To evaluate whether seven days of mifepristone treatment will result in a durable change in symptoms persisting after active treatment discontinuation, as measured by Borderline Personality Disorder Severity Index (BPDSI) total score. The BPDSI is a semi-structured clinical interview assessing the frequency and severity of manifestations of Borderline Personality Disorder (BPD) during a circumscribed period of the previous 7 days. The BPDSI measures 9 symptoms associated with BPD on a Likert scale ranging from 0-7 (0 = never; 7 = daily). Each symptom measure produces a mean score ranging from 0-7, with a higher score indicating more prevalent symptoms. A total score is then calculated using the summed symptom mean scores, ranging from 0-63, with a higher score indicating more prevalent symptoms.
Time Frame: 7 days of study medication to 21 days after discontinuation of study medication
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  BPDSI Total Score after 7 days of medication | 13.50 (7.93) | 9.45 (4.24)
  BPDSI Total Score 21 days after discont. study med | 13.58 (5.31) | 8.17 (4.32)

3. Primary Outcome: Number of Participants With Possibly and Probably Related Adverse Events
Description: To determine the safety and tolerability of mifepristone according to subject report of possibly and probably related adverse events (AEs). AEs were evaluated by study physicians at each visit and each reported AE was evaluated for relatedness (unrelated, possibly related, or probably related) to the study drug/procedure.
Time Frame: Baseline to 21 days after discontinuation of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Participants
  Number of subjects with possibly related AEs | 9 | 6
  Number of subjects with probably related AEs | 3 | 3

4. Primary Outcome: Levels of Cortisol
Description: To assess cortisol levels as a potential biomarker of hypothalamic-pituitary-adrenal (HPA)-axis engagement
Time Frame: Baseline (Visit 2), 7 days of study medication (Visit 4), 7 days after discontinuation of study medication (Visit 5), 21 days after discontinuation of study medication (Visit 6)
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
mcg/dL
  Cortisol Level - Baseline | 13.88 (5.39) | 14.38 (8.58)
  Cortisol Level - 7 days of study med | 35.01 (17.41) | 16.33 (9.50)
  Cortisol Level - 7 days after disc of study med | 20.91 (5.53) | 14.30 (6.88)
  Cortisol Level - 21 days after disc study med | 11.90 (4.95) | 15.73 (12.00)

5. Secondary Outcome: Symptom Change - BPDSI Subscales
Description: Borderline Personality Disorder Severity Index (BPDSI) symptom domain subscales scores. The BPDSI is a semi-structured clinical interview assessing the frequency and severity of manifestations of Borderline Personality Disorder (BPD) during a circumscribed period of the previous 7 days. The BPDSI measures 9 symptoms associated with BPD on a Likert scale ranging from 0-7 (0 = never; 7 = daily). Each symptom measure produces a mean score ranging from 0-7, with a higher score indicating more prevalent symptoms.
Time Frame: Baseline (Visit 2)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  BPDSI Subscale Score - Abandonment | 1.46 (0.96) | 1.36 (1.55)
  BPDSI Subscale Score - Interpersonal Relationships | 1.34 (0.91) | 0.70 (0.77)
  BPDSI Subscale Score - Identity | 2.76 (1.14) | 1.49 (1.34)
  BPDSI Subscale Score - Impulsivity | 0.78 (0.62) | 0.32 (0.37)
  BPDSI Subscale Score - Parasuicidal Behavior | 0.48 (0.62) | 0.30 (0.46)
  BPDSI Subscale Score - Affective Instability | 4.40 (1.79) | 4.48 (2.41)
  BPDSI Subscale Score - Emptiness | 3.96 (2.17) | 2.35 (1.39)
  BPDSI Subscale Score - Outbursts of Anger | 1.45 (1.27) | 1.53 (2.36)
  BPDSI Sub. Score-Dissociation & Paranoid Ideation | 1.45 (0.98) | 1.14 (1.28)

6. Secondary Outcome: Symptom Change - BPRS
Description: The Brief Psychiatric Rating Scale (BPRS) is an 19-item scale measuring positive symptoms, general psychopathology and affective symptoms during the last 7 days. The BPRS measures symptoms with scores ranging from 0-7, with a higher score indicating more severity. A total score is then calculated by adding all the item scores, ranging from 0-133, with a higher score indicating more severity.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  BPRS - Baseline | 37.70 (5.85) | 37.50 (7.09)
  BPRS - 7 days of study medication | 33.90 (6.15) | 33.36 (7.30)
  BPRS - 7 days after disc of study med | 35.78 (6.57) | 33.50 (7.66)
  BPRS - 21 days after disc study med | 35.22 (6.34) | 30.50 (5.44)

7. Secondary Outcome: Symptom Change - Borderline Checklist
Description: The Borderline Personality Checklist (BPD Checklist) is a 47-item DSM-IV based self-report questionnaire, designed to assess the experienced burden of specific BPD symptoms during the previous week. The BPD Checklist measures symptoms with scores ranging from 1-5, with a higher score indicating more severity. A total score is then calculated by adding all the item scores, ranging from 47-235, with a higher score indicating more severity.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  BPD Checklist - Baseline | 103.60 (30.83) | 96.92 (26.29)
  BPD Checklist - 7 days of study med | 98.10 (27.22) | 88.36 (32.02)
  BPD Checklist - 7 days after disc of study med | 91.56 (26.74) | 82.80 (37.94)
  BPD Checklist - 21 days after disc study med | 87.89 (24.31) | 78.80 (28.01)

8. Secondary Outcome: Symptom Change - SCL-90-R
Description: The Symptom Checklist-90-Revised (SCL-90-R) instrument helps evaluate a broad range of psychological problems and symptoms of psychopathology. The instrument is also useful in measuring patient progress or treatment outcomes. The SCL-90-R contains 90 items on a 5-point rating scale, with a higher score indicating more severity. The items are categorized into 12 domains (9 scores along primary symptom dimensions and 3 scores among global distress indices). A t-score for each domain is then obtained by norming by sex and ranges between 19-81, with a higher score indicating more severity.
Time Frame: Baseline (Visit 2)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  SCl-90-R - Somatization | 55.80 (6.18) | 50.25 (9.96)
  SCL-90-R - Obsessive-Complusive | 56.20 (8.48) | 51.50 (9.04)
  SCL-90-R - Interpersonal Sensitivity | 56.50 (12.19) | 51.58 (7.55)
  SCL-90-R - Depression | 54.40 (8.91) | 49.75 (9.20)
  SCL-90-R - Anxiety | 52.60 (9.09) | 47.17 (7.72)
  SCL-90-R - Hostility | 53.70 (8.54) | 53.00 (7.60)
  SCL-90-R - Phobic Anxiety | 50.00 (8.94) | 54.58 (11.05)
  SCL-90-R - Paranoid Ideation | 56.40 (9.75) | 48.45 (7.66)
  SCL-90-R - Psychoticism | 52.20 (9.37) | 47.67 (8.55)
  SCL-90-R - Global Severity Index | 55.20 (9.16) | 50.00 (8.42)
  SCL-90-R - Positive Symptom Total | 55.90 (10.72) | 49.00 (7.95)
  SCL-90-R - Positive Symptom Distress Index | 54.50 (7.49) | 52.25 (8.92)

9. Secondary Outcome: Metacognitive Capacity
Description: The Indiana Psychiatric Illness Interview (IPII) is a semi-structured interview developed to assess illness narratives. Responses are audio taped and later transcribed. It is scored using the Metacognition Assessment Scale- Abbreviated (MAS-A), which has four domains of metacognition: i) Self-Reflectivity ranging from 0-9; ii) Understanding the Mind of Other ranging from 0-7; iii) Decentration ranging from 0-3; and iv) Mastery ranging from 0-9. Lower scores indicate metacognitive deficits, higher scores indicate more integrated and nuanced metacognition. MAS-A total score is the sum of the scores on each of the domains of metacognition, ranging from 0-28, with a lower score indicating metacognitive deficits and a higher score indicating more integrated and nuanced metacognition.
Time Frame: Baseline, 21 days after discontinuation of study medication
Population: The IPII assessment was added to the study midway through the study therefore, the first 10 subjects did not have this assessments.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 6 | 6
Scores on a scale
  IIPI - Self-Reflectivity - Baseline | 5.08 (1.63) | 4.63 (1.70)
  IIPI-Self-Reflectivity-21 days after dis study med | 5.25 (1.89) | 3.90 (0.42)
  IIPI - Understanding Others - Baseline | 3.25 (1.08) | 2.88 (1.31)
  IIPI-Understanding Others-21 days after dis meds | 2.75 (0.50) | 2.50 (1.00)
  IIPI - Decentration - Baseline | 0.50 (0.45) | 0.38 (0.48)
  IIPI-Decentration-21 days after dis meds | 0.38 (0.75) | 0.20 (0.45)
  IIPI - Mastery - Baseline | 2.67 (1.89) | 3.88 (2.10)
  IIPI-Mastery-21 days after dis meds | 2.75 (0.50) | 2.80 (1.64)
  IIPI - Total - Baseline | 11.50 (4.69) | 11.75 (4.99)
  IIPI-Total-21 days after dis meds | 11.13 (2.95) | 9.40 (2.43)

10. Secondary Outcome: Symptom Change - CGI-S
Description: The Clinical Global Impressions Severity Scale (CGI-S) is used for repeated evaluations of global psychopathology. The CGI-S scale is widely used in schizophrenia research and is a single 7-point Likert scale rating severity of psychopathology on a scale of 1 (normal, not ill) to 7 (very severely ill), with a higher score indicating more severity.
Time Frame: Baseline, 7 days of study medication (Visit 4), 21 days after discontinuation of study medication (Visit 6)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  CGI-S - Baseline | 4.30 (0.67) | 4.42 (0.90)
  CGI-S - 7 days of study med | 4.20 (1.03) | 4.09 (1.04)
  CGI-S - 21 days after disc of study med | 3.89 (0.93) | 3.70 (0.95)

11. Secondary Outcome: Symptom Change - CGI-I
Description: The Clinical Global Impressions Improvement (CGI-I) scale is used to assess the clinical change as compared to symptoms at baseline using a 7-point Likert scale, ranging from very much improved (1) to very much worse (7), with a higher score indicating more severity.
Time Frame: 7 days of study medication (Visit 4), 21 days after discontinuation of study medication (Visit 6)
Population: The CGI-I is measured at visits after baseline, there was 1 subject taking Placebo who discontinued prior to Visit 4 and therefore was not included in analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 11
Scores on a scale
  CGI-I - 7 days of study med | 3.30 (1.16) | 3.36 (1.29)
  CGI-I - 21 days after disc of study med | 3.44 (1.01) | 2.80 (1.14)

12. Secondary Outcome: Symptom Change - BPDSI Subscales
Description: as for outcome 5
Time Frame: 7 days of study medication (Visit 4)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  BPDSI Subscale Score - Abandonment | 0.90 (0.59) | 1.27 (1.15)
  BPDSI Subscale Score - Interpersonal Relationships | 0.80 (0.54) | 0.58 (0.53)
  BPDSI Subscale Score - Identity | 1.64 (1.13) | 1.34 (0.85)
  BPDSI Subscale Score - Impulsivity | 0.66 (0.64) | 0.11 (0.17)
  BPDSI Subscale Score - Parasuicidal Behavior | 0.37 (0.52) | 0.19 (0.37)
  BPDSI Subscale Score - Affective Instability | 3.67 (2.43) | 2.89 (1.90)
  BPDSI Subscale Score - Emptiness | 2.76 (1.81) | 1.51 (0.91)
  BPDSI Subscale Score - Outbursts of Anger | 1.08 (1.20) | 0.79 (0.92)
  BPDSI Sub. Score-Dissociation & Paranoid Ideation | 1.63 (1.26) | 0.77 (0.84)

13. Secondary Outcome: Symptom Change - BPDSI Subscales
Description: as for outcome 5
Time Frame: 21 days after discontinuation of study medication (Visit 6)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  BPDSI Subscale Score - Abandonment | 1.06 (0.75) | 0.63 (0.67)
  BPDSI Subscale Score - Interpersonal Relationships | 0.84 (0.86) | 0.64 (0.88)
  BPDSI Subscale Score - Identity | 1.92 (1.12) | 0.63 (0.76)
  BPDSI Subscale Score - Impulsivity | 0.53 (0.58) | 0.11 (0.14)
  BPDSI Subscale Score - Parasuicidal Behavior | 0.43 (0.38) | 0.25 (0.37)
  BPDSI Subscale Score - Affective Instability | 3.27 (2.10) | 2.96 (1.60)
  BPDSI Subscale Score - Emptiness | 2.94 (1.86) | 1.79 (1.67)
  BPDSI Subscale Score - Outbursts of Anger | 0.97 (1.22) | 0.62 (1.07)
  BPDSI Sub. Score-Dissociation & Paranoid Ideation | 1.62 (1.03) | 0.56 (0.58)

14. Secondary Outcome: Symptom Change - SCL-90-R
Description: as for outcome 8
Time Frame: 7 days of study medication (Visit 4)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  SCl-90-R - Somatization | 53.00 (10.92) | 46.27 (9.18)
  SCL-90-R - Obsessive-Complusive | 54.30 (11.49) | 47.91 (9.69)
  SCL-90-R - Interpersonal Sensitivity | 53.00 (10.07) | 48.45 (10.05)
  SCL-90-R - Depression | 52.60 (9.32) | 47.82 (10.05)
  SCL-90-R - Anxiety | 49.10 (10.08) | 43.09 (9.39)
  SCL-90-R - Hostility | 52.80 (9.07) | 52.00 (10.85)
  SCL-90-R - Phobic Anxiety | 49.60 (6.59) | 49.55 (7.88)
  SCL-90-R - Paranoid Ideation | 53.80 (10.38) | 47.91 (8.88)
  SCL-90-R - Psychoticism | 48.80 (8.16) | 47.27 (10.67)
  SCL-90-R - Global Severity Index | 52.30 (9.89) | 45.82 (9.29)
  SCL-90-R - Positive Symptom Total | 53.40 (11.89) | 46.91 (9.69)
  SCL-90-R - Positive Symptom Distress Index | 54.20 (11.49) | 51.91 (17.04)

15. Secondary Outcome: Symptom Change - SCL-90-R
Description: as for outcome 8
Time Frame: 21 days after discontinuation of study medication (Visit 6)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 10 | 12
Scores on a scale
  SCl-90-R - Somatization | 49.78 (15.21) | 47.60 (10.70)
  SCL-90-R - Obsessive-Complusive | 51.33 (9.80) | 44.60 (12.69)
  SCL-90-R - Interpersonal Sensitivity | 48.89 (10.48) | 45.30 (8.79)
  SCL-90-R - Depression | 49.00 (9.86) | 44.00 (12.44)
  SCL-90-R - Anxiety | 48.44 (9.25) | 42.70 (10.27)
  SCL-90-R - Hostility | 50.11 (12.50) | 48.80 (6.84)
  SCL-90-R - Phobic Anxiety | 46.00 (6.96) | 50.10 (8.75)
  SCL-90-R - Paranoid Ideation | 50.33 (10.48) | 46.80 (12.56)
  SCL-90-R - Psychoticism | 45.44 (8.50) | 45.70 (13.31)
  SCL-90-R - Global Severity Index | 49.00 (10.30) | 45.10 (12.05)
  SCL-90-R - Positive Symptom Total | 49.56 (11.22) | 44.80 (10.40)
  SCL-90-R - Positive Symptom Distress Index | 51.67 (13.19) | 46.60 (12.47)

ADVERSE EVENTS:
Time Frame: Screening through 21 days after study medication was discontinued
Arm/Group | Mifepristone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/12
Other Adverse Events (participants affected / at risk) | 10/10 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=10) | Placebo (N=12)
Foreign body in urethra (Renal and urinary disorders) | 0 (0) | 1 (1) — Hospitalization for a foreign body in the urethra
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=10) | Placebo (N=12)
Abnormal electrocardiogram (Cardiac disorders) | 2 (2) | 1 (1)
Abdominal bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 2 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Atopic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blurry Vision (Eye disorders) | 2 (2) | 0 (0)
Bug Bites (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cramping (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Decreased Appetite (General disorders) | 0 (0) | 1 (1)
Decreased Concentration (General disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dizziness (General disorders) | 1 (1) | 0 (0)
Dog Bite Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry Eyes (Eye disorders) | 1 (1) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Exacerbation of borderline personality disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Exhaustion (General disorders) | 1 (1) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hand tremor (General disorders) | 1 (1) | 1 (1)
Headache/migraine (General disorders) | 3 (3) | 4 (4)
Heaviness in legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hemorrhoids (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Increased appetite (General disorders) | 0 (0) | 1 (1)
influenza (General disorders) | 0 (0) | 1 (1)
insomnia (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 2 (2)
lactation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
lump in throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
menstural bleeding (Reproductive system and breast disorders) | 1 (1) | 1 (2)
mouth sores (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pre-existing restless leg syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shakiness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sinus congestion (General disorders) | 1 (1) | 0 (0)
Somnolence (General disorders) | 3 (3) | 0 (0)
Toothache (General disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 3 (3)
worsening acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT01212588/Prot_SAP_000.pdf